CLINICAL TRIAL: NCT07154238
Title: Characteristics and Treatment Experiences of Individuals Using Injectable Semaglutide for Weight Management, a Cross-sectional Time-series Analysis, Multi-country Study.
Acronym: OUTSTEP-1
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN9536-8412; U1111-1314-6149 (Other: WHO)
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Baseline: 0 - 8 weeks post-initiation, individuals who self-reported an initiation date as day, month and year combination that is no more than eight weeks prior to the date that they complete the screener to participate in the study.
  Interventions: Other: No treatment given
- End of Escalation Phase: 16 - 24 weeks post-initiation, individuals who self-reported an initiation date as day, month and year combination that is at least 16 weeks but no more than 24 weeks prior to the date that they complete the screener to participate in the study.
  Interventions: Other: No treatment given
- Weight Loss Phase: 48 - 56 weeks post-initiation, individuals who self-reported an initiation date as day, month and year combination that is at least 48 weeks but no more than 56 weeks prior to the date that they complete the screener to participate in the study
  Interventions: Other: No treatment given
- Stable Weight Phase: More than or equal to (≥) 68 weeks post-initiation, individuals who self-reported an initiation date as day, month and year combination that is at least 68 weeks prior to the date that they complete the screener to participate in the study.
  Interventions: Other: No treatment given
- Healthcare Providers (HCP)s: HCPs will be recruited from an opt-in panel available in each country which includes the practitioners representing different settings of obesity care. Qualified HCPs will be invited to participate in a one-on-one IDI with a moderator from each of the participating countries.
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this study is to collect information for scientific research and to better understand the experiences of participants managing their weight. The study aims to collect valid responses through online interviews from participants. This study is a survey-based study without collection of laboratory data. Duration of the study will be about 14 months.

ELIGIBILITY:
Inclusion Criteria:

* For an eligible participant (individuals initiated on injectable semaglutide for weight management), all inclusion criteria must be answered "yes".

  1. Electronically provided consent obtained before any study-related activities can be completed.
  2. Age above or equal to 18 years at the time of providing informed consent.
  3. Reside in a participating country: Australia, Germany, United Arab Emirates (UAE) and Spain.
  4. Have been prescribed and initiated injectable semaglutide for weight management prior to study screening.
* For an eligible participant (HCPs), all inclusion criteria must be answered "yes".

  1. Electronically provided consent obtained before any study-related activities can be completed.
  2. Practice in a participating country: Australia, Germany, UAE, and Spain.
  3. See at least 150 patients for any condition per month; priority given to those who treat at least 200 patients for any condition per month.
  4. Treat at least 10 adult patients per month for weight management.
  5. Prescribe anti-obesity medications (AOMs) to their patients they personally treat for weight management/obesity care; priority given to those who treat at least 10% of the patients they personally treat for weight management/obesity care with anti-obesity medications (AOMs).
  6. Prescribe injectable semaglutide for weight management.
  7. Be a specialty of interest (varies by country); mix of primary care, specialists such as Endocrinologists, Diabetologists, Nutrition Specialists, Obesity Specialists and others.

Exclusion Criteria:

* For an eligible participant (individuals initiated on injectable semaglutide for weight management), all exclusion criteria must be answered "no".

  1. Unwillingness or language barriers precluding adequate understanding or cooperation.
  2. Is currently or planning to become pregnant in next six months.
  3. Is taking injectable semaglutide for Type 2 diabetes management only.
* For an eligible participant (HCPs), all exclusion criteria must be answered "no".

  1. Prior participation in this study. Participation is defined as having given informed consent and submitting responses to an interview.
  2. Unwillingness or language barriers precluding adequate understanding or cooperation.
  3. Only treats patients under 18 years of age.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will collect quantitative and qualitative data from individuals treated with injectable semaglutide for weight management in real-world settings.
  The study will include two groups of participants:
  1. Individuals who belong to or are recruited to an opt-in panel in the countries of interest and who have initiated injectable semaglutide for weight management. They will be classified according to the time when they first initiated treatment with injectable semaglutide for weight management.
  2. HCPs who prescribe injectable semaglutide for weight management will be recruited from an existing opt-in panel in the countries of interest.
Sampling Method: Non-Probability Sample
Enrollment: 2546 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Description of characteristics, including clinical, demographic and physical characteristics, among individuals initiated on injectable semaglutide for weight management | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list Single select from a defined list Numeric entry Open-ended type-in Patient Qualitative Segment Open-ended commentary
Description of the experience of individuals initiated on injectable semaglutide for weight management through personal perception of physical and mental health and self-reported QoL | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates extremely dissatisfied and 7 indicates extremely satisfied) Single select from a defined list EQ-5D-5L Patient Qualitative Segment Open-ended commentary
Individual-reported change in BMI since initiation | At the time of survey response (Day 1)
  Patient Quantitative Segment Numeric entry (BMI calculated based on self-reported height and weight)
Individual-reported achievement of weight loss goal | At the time of survey response (Day 1)
  Patient Quantitative Segment Yes/No; percentage of weight loss goal achieved Patient Qualitative Segment Open-ended commentary
Individual-reported change in weight since initiation | At the time of survey response (Day 1)
  Patient Quantitative Segment Numeric entry in (kgs); percentage of weight change Patient Qualitative Segment Open-ended commentary
Individual-reported changes in daily life since initiation on injectable semaglutide | At the time of survey response (Day 1)
  Patient Qualitative Segment Open-ended commentary

SECONDARY OUTCOMES:
Treatment expectation of individuals initiated on injectable semaglutide of ability to achieve weight loss goal using injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates not at all confident and 7 indicates extremely confident) Patient Qualitative Segment Open-ended commentary
Expectation for length of time of treatment to desired result from date of initiation on injectable semaglutide at baseline | At the time of survey response (Day 1)
  Patient Quantitative Segment Numeric entry months Patient Qualitative Segment Open-ended commentary
Expectation of individuals initiated on injectable semaglutide for weight management who believe they will have greater success in achieving their weight loss with the use of injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Patient Qualitative Segment Open-ended commentary
Expected benefits of injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list
Satisfaction with weight loss since initiation | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for satisfaction (where 1 indicates extremely dissatisfied all and 7 indicates extremely satisfied) Patient Qualitative Segment Open-ended commentary
Overall satisfaction with injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for satisfaction (where 1 indicates extremely dissatisfied all and 7 indicates extremely satisfied) Patient Qualitative Segment Open-ended commentary
Individual-reported changes in perception of injectable semaglutide since initiation | At the time of survey response (Day 1)
  Patient Qualitative Segment Open-ended commentary
Attitudes of individuals related to obesity or weight related stigmatization or discrimination prior to/since/due to initiation on injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list
Attitudes of individuals initiated on injectable semaglutide for weight management related to obesity as a chronic disease | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree)
Attitudes of individuals initiated on injectable semaglutide for weight management related to weight loss being their responsibility | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree)
Attitudes of individuals initiated on injectable semaglutide for weight management related to weight loss being more likely with use of prescription medication for weight loss (AOMs) | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree)
Degree of knowledge of individuals initiated on injectable semaglutide for weight management related to how prescription weight loss medications (AOMs) work in the body | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Patient Qualitative Segment Open-ended commentary
Behaviours of individuals initiated on injectable semaglutide for weight management related to making lifestyle changes in addition to initiating on injectable semaglutide for weight loss or weight management to achieve their weight loss goals | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Attitudes of individuals initiated injectable semaglutide for weight management related to the necessity to make lifestyle changes in addition to initiating injectable semaglutide for weight loss or weight management to achieve their weight loss goals | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Patient Qualitative Segment Open-ended commentary
Attitudes of individuals who initiated on injectable semaglutide for weight management relating to ease of maintaining lifestyle changes (e.g., eating a healthy diet and getting regular exercise) since initiating on injectable semaglutide | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree)
Individual-reported change in overall knowledge of how AOMs work from initiation on injectable semaglutide to present day | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree)
Attitudes related to viewing obesity as a chronic disease | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Attitudes related to belief weight loss is solely an individual's responsibility | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Attitudes related to belief weight loss requires use of prescription medication for weight loss (AOMs) | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Attitudes related to belief individuals must make lifestyle changes in addition to initiating on injectable semaglutide for weight loss or weight management to achieve their weight loss goals | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Attitudes related to belief individuals will have greater success in achieving their weight loss goals with use of injectable semaglutide | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Attitudes related to level of comfort prescribing AOMs and injectable semaglutide specifically for weight management | At the time of survey response (Day 1)
  HCP Qualitative Segment 7-point Likert scales for agreement (where 1 indicates strongly disagree and 7 indicates strongly agree) Open-ended commentary
Reasons for length of adherence | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Future planned use of injectable semaglutide (among current users) | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list; Numeric entry months Patient Qualitative Segment Open-ended commentary
Reasons for discontinuation (among those who discontinued) | At the time of survey response (Day 1)
  Patient Quantitative Segment Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Likelihood to resume injectable semaglutide (specifically for weight management) after formal discontinuation and reasons | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for likelihood (where 1 indicates not at all likely and 7 indicates extremely likely) Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Individual-reported likelihood of continuation on injectable semaglutide until achieve goal weight and reasons | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for likelihood (where 1 indicates not at all likely and 7 indicates extremely likely)
Likelihood of continuation on injectable semaglutide after achieving weight loss goal and reasons | At the time of survey response (Day 1)
  Patient Quantitative Segment 7-point Likert scale for likelihood (where 1 indicates not at all likely and 7 indicates extremely likely)
Treatment pause initiated by individual and reasons | At the time of survey response (Day 1)
  Patient Quantitative Segment Yes/No; Numeric entry; Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Treatment pause initiated by HCP and reasons | At the time of survey response (Day 1)
  Patient Quantitative Segment Yes/No; Numeric entry; Multi select from a defined list Patient Qualitative Segment Open-ended commentary
Number of treatment pauses | At the time of survey response (Day 1)
  Patient Quantitative Segment Numeric entry
Among those with low likelihood to use injectable semaglutide after discontinuation, potential use of another AOM | At the time of survey response (Day 1)
  Patient Quantitative Segment Yes/No/Not Sure

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bad Oeynhausen, Germany

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: https://novonordisk-trials.com